CLINICAL TRIAL: NCT03802370
Title: Soft Tissue Augmentation Using The Dome Technique Around Immediate Implants In The Esthetic Zone. A Case Series
Brief Title: Soft Tissue Augmentation Around Immediate Implants In The Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Abbas Elsayed, professor: Mona Shoeib , associated professor: Enji ahmed mahmoud, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-01-10
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: single arm groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single am (Other): single arm , superiority trial , tunneling technique in connective tissue graft around dental implants
  Interventions: Procedure: connective tissue grafting by Dome Technique

INTERVENTIONS:
Procedure: connective tissue grafting by Dome Technique — The dome technique addresses the placement of the CT, as it is layered over the implant and takes the shape of an inverted dome
  Other Names: Dome technique

SUMMARY:
Following tooth loss, a considerable reduction in hard- and soft-tissue volume can be expected (Tan WL, et al., 2012), (AraujoMG, et al., 2015). In the anterior maxilla, tissue loss can make future implant restorations more challenging and less predictable in terms of achieving and maintaining favorable soft-tissue-emergence profiles. Even with careful implant planning and placement, marginal gingival recession of 0.5-1 mm has been a common finding with single-tooth implants (Nisapakultorn K, et al., 2010), (Suphanantachat S, et al., 2012). This is partly attributed to bone remodeling after implant surgery, and occurs regardless of implant-placement protocol used (Hof M, et al., 2015).

DETAILED DESCRIPTION:
The dome technique addresses the placement of the CT, as it is layered over the implant and takes the shape of an inverted dome. The advantage of the dome CT technique is that it allows for both buccal and coronal augmentation of local soft tissue, while maximizing blood supply to the area by using tunneling-technique principles. It enhances and augments the peri-implant tissue foundation for a favorable facial and interproximal restorative emergence profile. As this technique does not involve raising an independent buccal flap, the gingival tissue of the adjacent teeth is not compromised, and thus the risk of recession and formation of black triangles on the adjacent teeth is minimized.

ELIGIBILITY:
Inclusion Criteria:

* Patients with healthy systemic condition
* Patients aged from 20 to 45 years old Availability of bone apical and palatal to the socket to provide primary stability.
* Presence of adequate gingival architecture with the surrounding dentition
* Patient provides an informed consent
* Adequate Inter-arch space for implant placement
* Favorable occlusion (no traumatic occlusion)
* Good oral hygiene
* Accepts 6-month follow-up period

Exclusion Criteria:

* Patients with signs of acute infection related to the area of interest
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as para-functional habits
* Current and former smokers
* Pregnant females
* HIV or Hepatitis; 5/Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Alcoholism or chronic drug abuse; 7/ Heavy smokers >10/cigarettes per day

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Pink esthetic score (PES) | 6 months
  The PES is based on seven variables mesial papilla, distal papilla, soft - tissue level, soft tissue contour, alveolar process deficiency, soft tissue color and texture . The PES is based on seven variables mesial papilla, distal papilla, soft - tissue level, soft tissue contour, alveolar process deficiency, soft tissue color and texture . it's numerical

SECONDARY OUTCOMES:
Gingival Thickness | 6 months
  Will be measured using an anesthetic needle with a rubber stopper, trans-gingivally piercing tissues horizontally perpendicular to the long axis of the tooth implant until it contacts bone
Post - Surgical Patient Satisfaction | 6 months
  A 3 - item questionnaire is asked and the patients shall use a 7point answer scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Irinakis T, Aldahlawi S. The dome technique: a new surgical technique to enhance soft-tissue margins and emergence profiles around implants placed in the esthetic zone. Clin Cosmet Investig Dent. 2018 Feb 14;10:1-7. doi: 10.2147/CCIDE.S154152. eCollection 2018. PMID 29491722